CLINICAL TRIAL: NCT00663130
Title: A Randomised, Double-blind, Double-dummy, Parallel-group, Active-controlled Study Evaluating the Efficacy of Vardenafil Versus Tadalafil When Intercourse is Attempted Within 45 Minutes of Administration in Subjects With Erectile Dysfunction
Brief Title: Evaluating the Efficacy Vardenafil 10 mg vs Tadalafil 10 mg in in Subjects With Erectile Dysfunction (ED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11333
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Active Comparator)
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Vardenafil 10mg, taken orally within 1 hour prior to sexual intercourse
  Arms: Arm 1
Drug: Tadalafil — Tadalafil 10mg, taken orally within 1 hour prior to sexual intercourse
  Arms: Arm 2

SUMMARY:
Evaluating the efficacy of 10mg vardenafil versus 10mg tadalafil in the first 45 minutes post-dosing, in an as-required regimen for 4 weeks in subjects with mild/moderate to severe ED

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 64 years
* Heterosexual males
* Erectile dysfunction for more than 6 months

Exclusion Criteria:

* Penile anatomical abnormalities
* Spinal cord injury
* History of surgical prostatectomy

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 759 (Actual)
Dates: Start 2004-04; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Sexual Encounter Profile Question 3 (SEP-3) | 4 weeks

SECONDARY OUTCOMES:
Sexual Encounter Profile Question 2 (SEP-2) | 4 weeks
International Index of Erectile Function | 4 weeks
Global Confidence Question (GCQ) | 4 weeks
Erection Quality Scale (EQS) | 4 weeks
General Safety | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer